CLINICAL TRIAL: NCT06997939
Title: A Clinical Trial of Autologous Bone Marrow-Derived Mesenchymal Stem Cell Transplantation for Precision Therapy in Ischemic Stroke
Brief Title: Autologous Bone Marrow Mesenchymal Stem Cell Therapy for Ischemic Stroke
Acronym: ABMSC-IS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Nantong Shengyuan Stem Cell Techology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-G097
Record Dates: First submitted 2025-05-18; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke
Keywords: autologous; bone marrow mesenchymal stem cell; mRS; functional recovery; Carotid artery intervention; NIHSS
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Single-center, three-arm parallel randomized controlled trial: Group A (Ommaya reservoir delivery), Group B (low-dose intra-arterial transplantation), and Group C (High-dose intra-arterial transplantation), with double-blinding.
Who Masked: Participant, Investigator
Masking Description: Double-blind design: Participants and investigators are masked to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ommaya Reservoir Group (Experimental): Stem Cell via Ommaya；2*10^7 cells dose
  Interventions: Biological: ABMSC
- Low-Dose intra-arterial transplantation group (Experimental): Internal carotid artery(ICA) transplantation；Low-dose; 2.5*10^6 cells dose
  Interventions: Biological: ABMSC
- High-Dose intra-arterial transplantation group (Experimental): Internal carotid artery(ICA) transplantation；High-dose; 1.0*10^7 cells dose
  Interventions: Biological: ABMSC

INTERVENTIONS:
Biological: ABMSC — Autologous bone marrow-derived mesenchymal stem cells administered via Ommaya reservoir；2.0*10^7 cell/dose
  Arms: Ommaya Reservoir Group
Biological: ABMSC — Autologous bone marrow-derived mesenchymal stem cells via intra-arterial route；Low-dose group; 2.5*10^6 cell/dose
  Arms: Low-Dose intra-arterial transplantation group
Biological: ABMSC — Autologous bone marrow-derived mesenchymal stem cells via intra-arterial route；High-dose group; 1.0*10^7 cell/dose
  Arms: High-Dose intra-arterial transplantation group

SUMMARY:
Stroke is a group of diseases mainly characterized by cerebral ischemia or hemorrhage, with a high fatality rate and disability rate. It has now become a major obstacle to social and economic development. Stem cells are a type of primitive cells with self-renewal, proliferation and differentiation potential. Under certain conditions, they can differentiate into cells of various tissues and organs. They have now become one of the key research directions for the repair of functional disorders after ischemic stroke. Compared with other types of stem cells, bone marrow mesenchymal stem cells (BMSCs) have the advantages of being relatively easy to obtain with less tissue damage, convenient and rapid in vitro expansion and culture, and the ability to actively migrate to the lesion area after injection without the risk of canceration.

This study plans to recruit and screen 12 subjects with ischemic stroke, divided into three groups (Ommaya drug reservoir group, low-dose internal carotid artery transplantation group, and high-dose internal carotid artery transplantation group), with 4 subjects in each group, for a clinical study of ABMSCs treatment for functional disorders after ischemic stroke. In accordance with the established treatment protocol, bone marrow will be collected from subjects during the stable phase of their condition, and ABMSCs will be infused three times via Ommaya drug reservoir/internal carotid artery within 1-6 months after collection. The study will assess the improvement of motor function in patients and analyze the feasibility and effectiveness of this therapy, laying a solid foundation for future clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years, both male and female
* Confirmed diagnosis of ischemic stroke within 3-12 months before enrollment.
* Moderate stroke with NIHSS score 5-12 at screening
* Modified Rankin Scale (mRS) score 3-5 (moderate to severe disability)
* Patient or legal guardian willing to provide written informed consent for treatment and study participation
* Able to comply with medical history collection, data storage, and follow-up procedures

Exclusion Criteria:

* Patients with needle phobia or lumbar spine disease affecting bone marrow aspiration
* Any acute illness at the time of screening
* Severe disability or end-stage disease
* Severe heart, liver, or kidney dysfunction
* Pulmonary infection or severe systemic infection
* History of severe allergic reactions
* Use of immunosuppressive drugs (e.g., steroids) within 3 months or vaccination within 6 months
* Any organic lesions causing increased intracranial pressure
* Current or past malignancy
* Seropositive for HIV, syphilis, hepatitis B, hepatitis C, or other severe infectious diseases
* Severe mental illness or impaired consciousness
* Coagulopathy or ongoing anticoagulant therapy
* Blood pressure ≥180/110 mmHg despite treatment
* Poorly controlled diabetes with advanced complications and Pre-existing conditions affecting limb mobility (e.g., claudication, osteoarthritis, rheumatoid arthritis, gouty arthritis)
* Participation in another clinical trial within 3 months
* Major surgery or trauma (including fractures) within 1 month
* Any other condition deemed unsuitable for study participation by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | 3-7 days post each transplantation and 6-month follow-up
  To assess safety, the number of AEs or SAEs will be evaluated

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale（NIHSS） score | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment and observation period and follow-up period compared with those before treatment
Modified Rankin Scale(mRS) score | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment, observation period and follow-up period compared with those before treatment
Modified Barthel Index | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment, observation period and follow-up period compared with those before treatment
Fugl-Meyer Assessment | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment, observation period and follow-up period compared with those before treatment
Fugl-Meyer Balance Assessment | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment, observation period and follow-up period compared with those before treatment
10-Meter Walk Test(10MWT) Time | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment, observation period and follow-up period compared with those before treatment
Functional Ambulation Category(FAC) | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment, observation period and follow-up period compared with those before treatment
Cerebral infarct volume changes on MRI | 6-month follow-up
  The changes during the follow-up period compared with those before treatment
Surface electromyography(sEMG) signal changes | 3-7 days post each transplantation and 6-month follow-up
  The changes during the treatment, observation period and follow-up period compared with those before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qiuhong Ji, MD, PhD, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No